CLINICAL TRIAL: NCT06732986
Title: Does the Structure of the Tendon Relate to the Temporal, Kinetic and Kinematic Jump Variables? Athletes Vs. Non Athletes: an Observational Study
Brief Title: Does the Structure of the Tendon Relate to the Temporal, Kinetic and Kinematic Jump Variables? Athletes Vs. Non Athletes
Status: Active, not recruiting | Type: Observational
Sponsor: Escola Superior de Tecnologia da Saúde do Porto (Other)
Responsible Party: Principal Investigator, Daniela Ferreira Carneiro, Master's degree in Physiotherapy, Escola Superior de Tecnologia da Saúde do Porto
Other Study IDs: CE0112D
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Vertical Jump; Patellar Tendon; Achilles Tendon
Keywords: Vertical jump; Jump performance; Patellar tendon; Tendon structure; UTC; Achilles tendon

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Athletes: The participants in the athlete group were volleyball players competing in the 1st or 2nd division of the Portuguese National Championship, training and/or competing for more than 20 hours per week.
- Non Athletes: The participants in the non-athlete group had no prior experience in any jumping sport.

SUMMARY:
The goal of this observational study is to investigate the relationship between temporal, kinetic, and kinematic jump variables and patellar and Achilles tendons' structure in athletes and non-athletes. The main research questions are:

Does the structure of the patellar and Achilles tendons relate to the temporal, kinetic, and kinematic jump variables? Does the relationship between these variables differ between athletes and non-athletes? To answer these questions, researchers will compare the two groups to determine if the relationships between the variables are similar. Participants will undergo a UTC (Ultrasound Tissue Characterization) scan of the patellar and Achilles tendons and perform five jumps: a countermovement jump, a single-leg countermovement jump on each leg and a single-leg horizontal jump on each leg.

ELIGIBILITY:
Inclusion Criteria for the Athletes Group:

1. Being a volleyball athlete competing in the 1st or 2nd division of the portuguese national championship;
2. Participating in training and games for more than 20 hours per week.

Exclusion Criteria for the Athletes Group:

1. Presence of any musculoskeletal, neurological, cardiorespiratory, or metabolic condition that affects jumping performance;
2. Absence from competition due to injury or illness in the last two weeks;
3. History of tendon rupture;
4. Previous tendon surgery;
5. Diagnosis of patellar tendinopathy in the last 12 months.

Exclusion Criteria for the Non-Athletes Group:

1. Presence of any musculoskeletal, neurological, cardiorespiratory, or metabolic condition that affects jumping performance;
2. Absence from competition due to injury or illness in the last two weeks;
3. History of tendon rupture;
4. Previous tendon surgery;
5. Diagnosis of patellar tendinopathy in the last 12 months;
6. Previous participation in a jumping sport.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The target population for this study consisted of young adults aged 18 to 35, of both sexes, including volleyball athletes and non-athletes.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Tendon Structure | Baseline
  Ultrasound Tissue Characterization (UTC) captures tendon structure and quantifies the number of altered fibers. This technology classifies tendon structure into four echo types, reflecting tendon integrity and fibrillar organization. Data collection for the patellar tendon will be conducted with participants seated, hips and knees at 90° flexion, and feet supported on a stable surface. For the Achilles tendon, the participants will be lying down with ankle in neutral position.
  This positioning ensures the probe is aligned transversely to the tendons, enabling the acquisition of optimal ultrasound images without anisotropy.
  Ultrasound parameters will be standardized for all scans: a 40-second B-mode ultrasound using a 7-10 Hz linear transducer, with the probe attached to a tracking device that moves automatically along the tendon's perpendicular axis, capturing consecutive images at 0.2 mm intervals. A single scan of the tendons will be performed for each knee.
Jump Variables | Baseline
  The data collection protocol includes the following tasks: countermovement jump, single-leg countermovement jump with the dominant leg, single-leg countermovement jump with the jumping leg, single-leg horizontal jump with the jumping leg and single-leg horizontal jump with the dominant leg. Kinematic variables will be analyzed by recording the spatial positions of reflective markers placed on specific anatomical regions. Data will be captured using the Qualisys Motion Capture System (version 2021.2).
  Ground reaction forces will be measured using a force platform connected to a signal amplifier. The platform records the three components of ground reaction forces-anteroposterior, mediolateral, and vertical-via four sensors.
  The image capture hardware is connected to the Qualisys USB Analog Acquisition interface, synchronizing temporal, kinetic, and kinematic data with the Qualisys Track Manager (QTM) software.

CONTACTS AND LOCATIONS:
Locations (1):
- Escola Superior de Saúde do Instituto Politécnico do Porto, Porto, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: No